CLINICAL TRIAL: NCT06740682
Title: The Effect of Potcost Stories on Childbirth Fear, Pain and Delivery Method
Brief Title: The Effect of Potcost Stories on Childbirth Fear,
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Mine Gokduman Keles, Dr, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2024/11 GO 2024/596
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Postnatal Care
Keywords: Potcost Stories; fear; pain; experiences; birth
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention)
- Potcost Stories (Active Comparator)
  Interventions: Behavioral: Podcast olumlu doğum hikayeler

INTERVENTIONS:
Behavioral: Podcast olumlu doğum hikayeler — ositive birth stories were listened to by women who gave birth in the hospital included in the study and created with their permission. The podcast recording was done in a single session. These positive birth stories were expertly reviewed by 3 obstetricians and 3 academics. Each podcast content is 10 to 20 minutes (Cai et al., 2023). A WhatsApp reminder msg will be sent so that the stories are not forgotten.
  In addition, the pregnant woman will be contacted by phone and trained to listen (Cai et al., 2023).
  Participants will be allowed to listen to the podcasts as much as they want (Cai et al., 2023). After listening to each story, their feedback will be received and the participants' doubts will be clarified. (Cai et al., 2023; Çankaya and Şimşek, 2021; Mousavi et al., 2022).
  Based on multimedia principles, podcast positive birth experiences will be prepared (Clark and Mayer, 2023). Week 24, Week 30-32, Week 36-38 First story
  Arms: Potcost Stories

SUMMARY:
Birth is an important period that affects a woman's life physically, psychologically and socially. Although this experience can bring joy, it can also be accompanied by anxiety and fear. Fear of birth is affected by people's past traumatic birth experiences, lack of information, and the transfer of birth experiences experienced by individuals . Birth stories are one of the most accessible and frequently used tools for women to learn about birth. These stories are seen to affect women's fears of birth and their birth preferences .This study will evaluate the impact of Potcost Stories on childbirth-related fear, pain, experiences and mode of delivery.

DETAILED DESCRIPTION:
Birth is an important period that affects a woman's life physically, psychologically and socially. Although this experience can bring joy, it can also be accompanied by anxiety and fear. Fear of birth is affected by people's past traumatic birth experiences, lack of information, and the transfer of birth experiences experienced by individuals . Birth stories are one of the most accessible and frequently used tools for women to learn about birth. These stories are seen to affect women's fears of birth and their birth preferences .The World Health Organization (WHO) has emphasized the importance of education given during pregnancy in reducing a positive birth experience and fear of birth. . Advances in technology have made podcasts, videos, and mobile phone applications (apps) widely used in training. As a result of these trainings, behavioral changes are observed in people. It has been reported that being supported by midwives during pregnancy and encouraging birth as a positive experience reduces the fear of birth . Therefore, sharing positive birth stories in pregnancy schools and antenatal care is of great importance. However, it is thought that using podcast stories and sharing women's positive birth experiences together will reduce fear during birth and increase vaginal birth. Therefore, in this study, a podcast of stories that pregnant women can listen to again whenever they want, including positive birth experiences, was prepared. This study aimed to determine the effects of potcost stories on fear, pain, satisfaction and birth outcomes related to birth. We aim for the findings and results of the study to contribute to the midwifery and nursing care literature.

This study will evaluate the effects of Potcost Stories on fear, pain, experiences and delivery type related to birth.

ELIGIBILITY:
Inclusion Criteria:

Those who have completed at least primary school education

* Those who can speak, understand and write Turkish
* Those between the ages of 18-35
* Those who have spontaneous pregnancy
* Those who volunteer to participate in the study
* Those who are in the 24th week of pregnancy according to their last menstrual period (LMT) or ultrasound (USG) records
* Those who have no risk factors
* Those who have a phone number that can be used for educational interviews
* Those who attend a pregnancy school

Exclusion Criteria:

* Those who have fear of childbirth

  * Those who have chronic and/or psychiatric health problems
  * Those who did not attend at least three sessions of the education program
  * Those who were at risk during the pregnancy at any stage of the study
  * Those who could not be interviewed within the first 24 hours after birth were excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Wijma Birth Expectation/Experience Scale (W-DEQ) Version A | 1 MOUNT
  The Wijma Birth Expectation/Experience Scale Version A (W-DEQ A), developed by K. Wijma et al. in Sweden in 1998, was adapted to Turkish by Körükçü et al. in 2012. The W-DEQ consists of 33 items and is a six-point Likert-type scale.
  The item responses are numbered from 0 to 5, with 0 indicating "completely" and 5 indicating "not at all". The minimum score that can be obtained from the scale is 0, and the maximum score is 165.
  The cut-off value is 85 points, and a score of 85 and above is expressed as clinical fear. A high total scale score means that the degree of fear experienced is also high.
  * W-DEQ score ? 37 is mild,
  * W-DEQ score = 38-65 is moderate,
  * W-DEQ score = 66-84 is severe,
  * W-DEQ score ? 85 indicates clinical fear. Questions 2, 3, 6, 7, 8, 11, 12, 15, 19, 20, 24, 25, 27 and 31 in the scale are negatively loaded and are calculated by reversing in order to ensure compliance in the measurement. The Cronbach a
VASA Pain | 1 HOUR
  The numerical pain rating scale (NAS) is used to assess pain intensity. In the numerical rating scale, pain is rated between 0 (absence of pain) and 10 (unbearable pain) (Price et al., 1983)
Birth Experience Questionnaire (CEQ) | 1 HOUR
  The Birth Experience Questionnaire (CEQ), developed by Dencker et al. in 2010, was adapted to Turkish by Mamuk et al. in 2019. The scale, which was developed to measure women's birth experience in different dimensions, has four sub-dimensions and 22 items. It consists of the Birth process with 8 items, Professional help / Support with 5 items, Perceived Security / Memories with 6 items and Participation in Decisions with 3 items.
  * Questions 1, 2, 4, 5, 6, 19, 20, 21 in the Birth Process sub-dimension;
  * Questions 13, 14, 15, 16, 17 in the Professional help / Support sub-dimension;
  * Questions 3, 7, 8, 9, 18, 22 in the Perceived Security / Memories sub-dimension;
  * Questions 10, 11, 12 are included in the Participation in Decisions sub-dimension.
  The first 19 items of the scale are in the four-point Likert type and are scored from 1 to 4.
  • Completely agree = 1, • Mostly agree = 2, • Partially agree = 3, • Strongly disagree = 4.
  The last three

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aslantas BN, Cankaya S. The effect of birth ball exercise on labor pain, delivery duration, birth comfort, and birth satisfaction: a randomized controlled study. Arch Gynecol Obstet. 2024 Jun;309(6):2459-2474. doi: 10.1007/s00404-023-07115-4. Epub 2023 Jul 5. PMID 37405439
- [Background] Alizadeh-Dibazari Z, Abdolalipour S, Mirghafourvand M. The effect of prenatal education on fear of childbirth, pain intensity during labour and childbirth experience: a scoping review using systematic approach and meta-analysis. BMC Pregnancy Childbirth. 2023 Jul 27;23(1):541. doi: 10.1186/s12884-023-05867-0. PMID 37501120
- [Background] Abadi Marzoni Z, Bakouei F, Aghajani Delavar M, Hamidia A, Sepidarkish M. Midwife-led psycho-education intervention to reduce childbirth fear: a quasi-experimental study. Health Educ Res. 2024 May 11;39(3):245-253. doi: 10.1093/her/cyae017. PMID 38687635